CLINICAL TRIAL: NCT04928092
Title: A Zero Acute Kidney Injury (Zero-AKI) Strategy for Percutaneous Coronary Intervention in Patients With ChronicKidney Disease
Brief Title: A Zero Acute Kidney Injury Strategy for Percutaneous Coronary Intervention in Patients With ChronicKidney Disease
Acronym: Zero-AKI
Status: Withdrawn | Type: Observational
Why Stopped: The PI is leaving the institution
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Guerbet (Industry)
Responsible Party: Sponsor
Other Study IDs: HM20019541
Record Dates: First submitted 2021-05-26; First posted 2021-06-16 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: Acute Kidney Injury; Coronary Artery Disease; Percutaneous Coronary Intervention
MeSH Terms: conditions — Acute Kidney Injury; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Active research group: Patients undergoing intravascular imaging guided, low contrast PCI procedure as part of standard care
  Interventions: Procedure: Standard of care Ultra Low Contrast PCI

INTERVENTIONS:
Procedure: Standard of care Ultra Low Contrast PCI — PCI using low amounts of contrast media which is standard of care at VCU Medical Center

SUMMARY:
The purpose of this study is to compare the outcomes of Percutaneous Coronary Intervention (PCI) in patients with chronic kidney disease (CKD) using smaller doses of contrast dye that are validated as being at low risk of causing injury to the kidneys, with the larger doses that are traditionally used contemporary practice.

DETAILED DESCRIPTION:
This study will evaluate whether using lower doses of contrast dye leads to lower rates of kidney injury compared to current standard of care. In particular, effort will be taken to maintain the total amount of contrast dye below a scientifically-validated threshold calculated on the basis of each participant renal function. Participants will already be scheduled to undergo a PCI. Because a smaller amount of contrast dye will be used, an intravascular ultrasound (IVUS) will be used to help the doctors see and open the blockages in participant's coronary arteries. IVUS is already used to optimize PCI results, but will be used more extensively in this case. The amount of contrast dye received will be tailored on each participant kidney function. Prospectively enrolled patients will be matched with historical controls who underwent PCI with non-intravascular imaging based approach.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients undergoing elective and urgent (i.e., non-emergent) PCI
* Age >18 years
* eGFR <60 ml/min/1.73 m2
* Angina or equivalent and/or documentation of inducible myocardial ischemia
* Presence of =1 coronary stenosis, evaluated >70% by visual estimation (on a previously performed coronary angiography) or with an FFR =0.80
* ability to provide written informed consent

Exclusion Criteria:

* Emergent PCI due to either hemodynamic instability, ST-elevation myocardial infarction or sudden cardiac death
* PCI on chronic total occlusion
* Prior PCI within 3 weeks
* Age >90 years
* Left ventricular ejection fraction <20%
* Need for mechanical circulatory support
* Pregnancy
* Prisoners
* Non-English speaking patients
* Inability to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled to undergo a PCI.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-01 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Acute Kidney Injury (AKI) | Up to 72 hours after the procedure
  Standard laboratory assays related to renal function will be used to identify which, if any, patients develop AKI

OTHER OUTCOMES:
Cardiac death | Up to 30 days after PCI procedure
  Number of cardiac deaths
Myocardial infarction | Up to 30 days after PCI procedure
  Number of myocardial infarctions
Target lesion revascularization | Up to 30 days after PCI procedure
  Number of target-lesion revascularizations
All-cause mortality | Up to 30 days after PCI procedure
  Number of deaths due to any cause
Pericardial effusion | Up to 30 days after PCI procedure
  Number of pericardial effusion
new need for dialysis | Up to 30 days after PCI procedure
  Number of new patients needing dialysis

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Azzalini, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No